CLINICAL TRIAL: NCT01432951
Title: Pharmacokinetics of Enzastaurin HCl in Native Chinese Patients With Advanced and/or Metastatic Solid Tumors or Lymphoma
Brief Title: A Study of Enzastaurin in Chinese Patients With Advanced and/or Metastatic Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13322; H6Q-FW-JCCC (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Results first posted 2020-09-02 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: Solid Tumor; Lymphoma, Malignant
MeSH Terms: conditions — Lymphoma | interventions — enzastaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enzastaurin (Experimental): Enzastaurin 500 mg, four 125-mg tablets administered orally once daily for 14 days. Dosing is held for 3 days, and resumes on Day 18. Participants may continue receiving optional enzastaurin for an additional 2 to 4 weeks.
  Safety Extension: Participants had the option to continue receiving enzastaurin until disease progression or discontinuation criteria are met, as per the investigator's assessment.
  Interventions: Drug: Enzastaurin

INTERVENTIONS:
Drug: Enzastaurin — Administered orally
  Other Names: LY317615

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK) of enzastaurin and its metabolites in native Chinese participants with advanced and/or metastatic solid tumors or lymphoma. Information about any side effects that may occur will also be collected. Treatment of disease is not the main purpose of the study.

This is a Phase 1 study of enzastaurin in native Chinese participants with advanced and/or metastatic solid tumors or lymphoma. Participants will receive daily doses of enzastaurin for 14 days, stop dosing for 3 days during PK sampling, and resume dosing on Day 18. Participants may be allowed to receive enzastaurin for approximately 2 to 4 weeks after day 18 to provide an opportunity for a participant's oncologist to assess the potential benefit of the participant continuing to receive enzastaurin in the safety extension phase. There is no planned duration for the extension phase; participants are allowed to continue receiving enzastaurin until disease progression or other reason for discontinuation as per the investigator's assessment.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Have a histologic or cytologic diagnosis of cancer (solid tumor or lymphoma) with clinical or radiologic evidence of locally advanced and/or metastatic disease for which no life-prolonging therapy exists. (Note: participants with glioblastoma, and other hematologic malignancies [except lymphoma] are excluded from this study.)
* Male and female participants with reproductive potential must use an approved contraceptive method, if appropriate (for example, intrauterine device, birth control pills, or barrier device) during and for 3 months after discontinuation of study treatment. Women with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.
* Have a performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) scale and, in the investigator's opinion, are suitable for participation in the study
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, anticancer hormone therapy, or other investigational therapy for at least 30 days prior to study entry (6 weeks for mitomycin-C or nitrosoureas), and have recovered from the acute effects of therapy
* If the participants have hormone-refractory prostate cancer, the study doctor will discuss with the participants what drugs they would be allowed to continue to receive during the study
* Have adequate organ function, including:

  * Bone Marrow Reserve: absolute neutrophil count (ANC) greater than or equal to 1.5 × 10^9/Liter (L) prior to treatment, platelets greater than or equal to 100 × 10^9/L, and hemoglobin greater than or equal to 10 gram/deciliter (g/dL). Participants may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Participants may be allowed erythropoietin of choice as per standard of care.
  * Hepatic: bilirubin within 1.5 times the upper limit of normal (ULN), alanine transaminase, and aspartate transaminase less than or equal to 2.5 times ULN or less than or equal to 5 times ULN when liver metastases are known
  * Renal: serum creatinine less than or equal to 1.5 milligram/deciliter (mg/dL)
* Electrolytes: Participants may be entered into the study if, in the investigator's opinion, any electrolyte disorders, including potassium less than 3.4 milliequivalents/liter (mEq/L), calcium less than 8.4 mg/dL, or magnesium less than 1.2 (mEq/L), may be appropriately managed and stabilized by the time of the laboratory evaluation on the lead-in day. If electrolytes have not been stabilized during this time, the participant will be discontinued from the study. Participants with hypercalcemia are excluded.
* Have an estimated life expectancy, in the judgment of the investigator, that will permit the participant to complete the PK phase and at least 1 cycle of the safety extension phase (if the participant were to participate in the safety extension phase)

Exclusion Criteria:

* Have received treatment within 28 days of the first dose of study drug with an experimental agent for non cancer indications that has not received regulatory approval for any indication
* Participants with glioblastoma or hematologic malignancies other than lymphoma are excluded from this study. Participants who have central nervous system (CNS) metastases (unless the participant has completed successful local therapy.

for CNS metastases and has been off of corticosteroids for at least 4 weeks before starting study therapy) are excluded. In the absence of a clinical suspicion of brain metastases, no screening computed tomography (CT) or magnetic resonance imaging (MRI) scan before enrollment is required.

* Serious concomitant systemic disorder, including active infection, that is incompatible with the study (at the discretion of the investigator)
* Have a history of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infections
* Have a serious cardiac condition
* Have abnormal electrocardiogram (ECG) findings, at the discretion of the investigator
* Use medications that are known to cause certain changes in electrocardiogram (ECG) readings
* Have a history of unexplained syncope (fainting or passing out) within the last year, or have a known family history of unexplained sudden death
* Have had a complete gastrectomy or other significant gastrointestinal diseases that, in the investigator's opinion, may significantly impact drug absorption
* Are receiving total parenteral nutrition
* Are not able to swallow tablets
* Are a woman who is breast feeding, lactating, or pregnant
* Are allergic to enzastaurin
* Are receiving herbal regimens
* Drugs and herbal supplements that are known to be potent or moderate inhibitors or inducers of cytochrome P450 (CYP)3A are specifically excluded. Foods that are known to be potent or moderate inhibitors of CYP3A (for example, grapefruit, grapefruit juice, Seville oranges, or Seville orange juice) are also specifically excluded during the study. In addition, starfruit and starfruit juice are excluded during the PK phase of the study.
* Drugs with narrow therapeutic windows that are also known substrates of CYP2C9, CYP2C8, CYP2C19, and CYP3A are excluded
* Have an average weekly alcohol intake that exceeds 21 units per week (men) and 14 units per week (women) or are unwilling to stop alcohol consumption from the lead-in day through the completion of collecting samples for study drug measurement (1 unit = 12 oz or 360 milliliter (mL) of beer; 5 ounces (oz) or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Use of drugs of abuse, as evidenced by history and/or positive findings on urinary drug screening, unless prescribed by a physician (for example, narcotic pain medication)
* The investigator thinks you should not participate for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01-11 (Actual); Study Completion 2018-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- China (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changsha
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou

REFERENCES:
- [Derived] Li X, Fang X, Li S, Zhang W, Yang N, Cui Y, Huang H, Cai R, Lin X, Fu X, Hong H, Lin T. A pharmacokinetic and safety study of a fixed oral dose of enzastaurin HCl in native Chinese patients with refractory solid tumors and lymphoma. Oncotarget. 2016 Apr 5;7(14):18585-93. doi: 10.18632/oncotarget.7875. PMID 26942463

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who were considered to have completed the study who received at least 1 dose of study drug and from whom a valid assay result was obtained.
Groups:
- Enzastaurin: Enzastaurin 500 mg, four 125-mg tablets was administered orally once daily for 14 days. Dosing is held for 3 days, and resumes on Day 18. Participants may continue receiving optional enzastaurin treatment for up to 30 days.
  Safety Extension: Participants had the option to continue receiving enzastaurin treatment until disease progression or discontinuation criteria are met, as per the investigator's assessment.
Period: Treatment Phase (Day 1 to 30)
Arm/Group | Enzastaurin
Started | 26
Received at Least One Dose of Study Drug | 25
PK Sampling (no Dosing) Days 15-17 | 23
Progressive Disease | 10
Completed | 25
Not Completed | 1
Not completed — Never Treated | 1
Period: Safety Extension Day 30 to End of Study
Arm/Group | Enzastaurin
Started | 15 (Participants had the option to continue on to safety extension period.)
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Enzastaurin: Enzastaurin 500 mg, four 125-mg tablets was administered orally once daily for 14 days. Dosing is held for 3 days, and resumes on Day 18. Participants may continue receiving optional enzastaurin treatment for up to 30 days.
Arm/Group | Enzastaurin
Number analyzed (Participants) | 26
Age, Continuous [Mean (Full Range); unit: years] | 52 [32 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 26
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 26

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration -Time Curve Over a Dosing Interval at Steady State (AUCt,ss) of Enzastaurin, It's Metabolites and Total Analytes in Plasma
Description: PK (AUCt,ss) of Enzastaurin, its metabolites (LSN326020, LSN485912, and LSN2406799), and total analyte in plasma (enzastaurin + LSN326020 + LSN485912 + LSN2406799) were reported.
Time Frame: Day 14: Predose and 1, 2, 4, 6, 8, 10, 24, 48, 72, and 96 hours post dose
Population: All participants who received at least one dose of study drug had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole*hour/Liter (nmol*h/L)
Arm/Group | Enzastaurin
Number analyzed (Participants) | 23
nanomole*hour/Liter (nmol*h/L)
  Enzastaurin | 29100 (128)
  LSN326020 | 21800 (45.5)
  LSN485912 | 6520 (145)
  LSN2406799 | 2910 (103)
  Total Analytes | 63700 (86.1)

2. Primary Outcome: PK: Maximum Observed Drug Concentration at Steady State (Cmax,ss) of Enzastaurin, It's Metabolites and Total Analytes in Plasma
Description: PK (Cmax,ss) of Enzastaurin, its metabolites (LSN326020, LSN485912, and LSN2406799), and total analyte in plasma (enzastaurin + LSN326020 + LSN485912 + LSN2406799) were reported.
Time Frame: Day 14: Predose and and 1, 2, 4, 6, 8, 10, 24, 48, 72, and 96 hours post dose
Population: All participants who received at least one dose of study drug had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/liter (nmol/L)
Arm/Group | Enzastaurin
Number analyzed (Participants) | 23
nanomole/liter (nmol/L)
  Enzastaurin | 2370 (112)
  LSN326020 | 1070 (38.4)
  LSN485912 | 385 (116)
  LSN2406799 | 265 (89.8)
  Total Analytes | 4140 (81.5)

3. Primary Outcome: PK: Time of Maximal Plasma Concentration at Steady State (Tmax, ss) of Enzastaurin, It's Metabolites and Total Analytes in Plasma
Description: PK (tmax,ss) of Enzastaurin, its metabolites (LSN326020, LSN485912, and LSN2406799), and total analyte in plasma (enzastaurin + LSN326020 + LSN485912 + LSN2406799) were reported.
Time Frame: Day 14: Predose and 1, 2, 4, 6, 8, 10, 24, 48, 72, and 96 hours post dose
Population: All participants who received at least one dose of study drug had evaluable PK data.
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Enzastaurin
Number analyzed (Participants) | 23
Hour (h)
  Enzastaurin | 4.00 [2.00 to 8.17]
  LSN326020 | 5.97 [0.00 to 24.00]
  LSN485912 | 6.00 [0.00 to 24.00]
  LSN2406799 | 4.00 [2.00 to 8.17]
  Total Analytes | 4.00 [2.00 to 8.17]

4. Primary Outcome: PK: Average Concentration During a Dosing Interval at Steady State (Cav,ss) of Enzastaurin, It's Metabolites and Total Analytes in Plasma
Description: PK (Cav,ss) of Enzastaurin, its metabolites (LSN326020, LSN485912, and LSN2406799), and total analyte in plasma (enzastaurin + LSN326020 + LSN485912 + LSN2406799) were reported.
Time Frame: Day 14: Predose and and 1, 2, 4, 6, 8, 10, 24, 48, 72, and 96 hours post dose
Population: All participants who received at least one dose of study drug had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Enzastaurin
Number analyzed (Participants) | 23
nmol/L
  Enzastaurin | 1210 (128)
  LSN326020 | 907 (45.5)
  LSN485912 | 272 (145)
  LSN2406799 | 121 (103)
  Total Analytes | 2650 (86.1)

5. Primary Outcome: PK: Terminal Elimination Half-Life of Enzastaurin, It's Metabolites and Total Analytes in Plasma
Description: PK terminal elimination half-life of Enzastaurin, its metabolites (LSN326020, LSN485912, and LSN2406799), and total analyte in plasma (enzastaurin + LSN326020 + LSN485912 + LSN2406799) were reported.
Time Frame: Day 14: Predose and 1, 2, 4, 6, 8, 10, 24, 48, 72, and 96 hours post dose
Population: All participants who received at least one dose of study drug had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour (h)
Arm/Group | Enzastaurin
Number analyzed (Participants) | 23
Hour (h)
  Enzastaurin | 14.0 (54.0)
  LSN326020 | 42.0 (42.2)
  LSN485912 | 14.5 (51.7)
  LSN2406799 | 15.4 (51.1)
  Total Analytes | NA (NA) — Total analytes are not directly measured or reported.

ADVERSE EVENTS:
Time Frame: From Baseline to Study Completion (Up to 6 years and 1 month)
Groups:
- Enzastaurin Safety Extension: Participants had the option to continue receiving enzastaurin 500 mg, orally once daily until disease progression or discontinuation criteria are met, as per the investigator's assessment.
Arm/Group | Enzastaurin | Enzastaurin Safety Extension
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/15
Other Adverse Events (participants affected / at risk) | 19/25 | 9/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin (N=25) | Enzastaurin Safety Extension (N=15)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 2 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (2)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Oedema (General disorders) | 1 (1) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (5)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 2 (2)
Blood bilirubin (Investigations) | 0 (0) | 1 (1)
Blood follicle stimulating hormone (Investigations) | 0 (0) | 1 (1)
Blood luteinising hormone increased (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram qt prolonged (Investigations) | 9 (11) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 4 (4)
Lymphocyte count decreased (Investigations) | 2 (2) | 1 (1)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Protein total decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days